CLINICAL TRIAL: NCT03621644
Title: Prospective Phase II Study of Stereotactic Magnetic Resonance Imaging (MRI) Guided On-table Adaptive Radiation Therapy (SMART) for Patients With Borderline or Inoperable Locally Advanced Pancreatic Cancer
Brief Title: Stereotactic MRI-guided On-table Adaptive Radiation Therapy (SMART) for Locally Advanced Pancreatic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Viewray Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VR C2T2 - SMART - LAPC/BRPC 1
Record Dates: First submitted 2018-07-26; First posted 2018-08-08 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Radiation Therapy; SBRT
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ablative MRIdian SMART (Experimental): Radiation: Stereotactic MRI-guided On-table Adaptive Radiation Therapy 50 Gy in 5 fractions
  Interventions: Radiation: Stereotactic MRI-guided On-table Adaptive Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic MRI-guided On-table Adaptive Radiation Therapy — Radiation therapy will be delivered with an integrated magnetic resonance imaging (MRI)-guided radiotherapy delivery system (ViewRay MRIdian or MRIdian Linac). The prescribed dose will be 50 Gray (Gy) in 5 fractions. Stereotactic body radiotherapy (SBRT) fractions will be delivered at least twice per week, and with at least 18 hours between fractions. Each participant will be aligned in the treatment system with MRI image-guidance. On-table adaptive re-planning will be used when clinically indicated. In all patients, real-time MRI imaging will be used throughout treatment delivery to monitor the target location and control the radiation beam as necessary.

SUMMARY:
High-dose magnetic resonance imaging (MRI) guided hypofractionated radiation therapy delivered using daily adaptive dose planning has been shown in a retrospective study to result in improved overall survival, relative to patients receiving lower radiation doses, in patients with locally advanced pancreatic cancer, without increasing the rate of serious gastrointestinal toxicity.

The goal of the proposed trial is to investigative in a controlled, prospective manner the robustness of this outcome, and to track quality of life over a 5-year trial period.

DETAILED DESCRIPTION:
Prior stereotactic body radiotherapy (SBRT) experiences for treatment of locally advanced pancreatic cancer entailed either single-fraction or multi-fraction approaches delivering 33 Gray (Gy) in 5 fractions. Excellent tolerance and tumor control has been demonstrated, but median survival remained approximately 14 months. This highlights the strengths and limitations of SBRT to current radiation doses for pancreatic cancer. A prior Washington University institutional study and retrospective review has shown the safety of delivering 67.5 Gy in 15 fractions for inoperable pancreatic cancer using a strict 'isotoxicity' approach of limiting the gastrointestinal (GI) organs at risk (stomach, duodenum, small bowel and large bowel) to 45 Gy to 0.5 cm3 or less. This regimen resulted in no grade 3 or higher GI toxicities, and only one death in the 19 patients with a median follow-up of 15 months. This is significantly improved from prior experiences, where approximately 15 months represents the median survival for most studies of inoperable pancreatic cancer.

A recent retrospective analysis of 42 locally advanced pancreatic cancer patients treated by magnetic resonance imaging (MRI) guided radiation therapy at four institutions (University of California, Los Angeles, University of Wisconsin, Vrije Universiteit Medical Center (VUmc), Amsterdam, and Washington University, St. Louis) demonstrated that high-dose stereotactic body radiotherapy (SBRT) or hypofractionated radiation therapy delivered using daily ADAPTIVE dose planning on an MRI-guided radiotherapy system (MRIdian, ViewRay Inc.) has the potential to further improve overall survival. A control group of 19 patients treated to more conventional radiation doses without frequent dose adaptation showed a median survival of 14.8 months, while patients treated to high radiation doses (n=23, maximum biologically equivalent dose at alpha/beta = 10 Gy, or BED10 of > 90 Gy) under daily or almost daily adaptive re-planning had an estimated median survival of 27.8 months (p=0.005). Interestingly, increased radiation dose delivery using daily dose adaptation was correlated with less grade 3 toxicity (0% in the high dose group vs 15.8% in patients treated to lower radiation doses without dose adaptation).

The compelling data of this retrospective study prompted the development of this current prospective clinical trial designed to assess the primary objective of grade 3 or greater GI toxicity at 90 days for patients with borderline resectable or inoperable locally advanced pancreatic cancer treated with MRI-guided on-table adaptive radiation therapy and soft tissue tracking with radiation beam gating to 50 Gy in 5 fractions. Secondary objectives include assessment of (1) overall survival at 2 years, (2) distant progression free survival at 6 months, and (3) changes in patient-reported quality of life (QOL) from pre-treatment to 3 and 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced adenocarcinoma of the pancreas that is considered unresectable or borderline resectable on institutional standardized criteria of unresectability or medical inoperability. Patients with and without regional adenopathy are eligible as long as lymph nodes are adjacent to primary tumor.
2. Greater than or equal to 3 months of systemic chemotherapy
3. At least 18 years of age.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
5. Normal bone marrow and organ function as defined below:

   1. Absolute neutrophil count ≥ 500/mcL (microliters)
   2. Platelets ≥ 50,000/mcL
   3. Hemoglobin ≥ 8.0 g/dL (deciliters)
   4. Total bilirubin ≤ 1.5 x IULN
   5. Aspartate Aminotransferase AST(SGOT) / Alanine Aminotransferase ALT(SGPT) ≤ 3.0 x Institutional Upper Limit of Normal (IULN)
6. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
7. Ability to understand and willingness to sign an Institutional Review Board (IRB) approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

1. Distant metastatic disease as assessed by staging positron emission tomography / computed tomography (PET/CT) or CT of the chest and abdomen within 6 weeks of starting radiation therapy
2. Carbohydrate antigen (CA19.9) > 500 U/ml.
3. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
4. Currently receiving any other investigational agents.
5. Major surgery within 4 weeks prior to first day of treatment.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
7. Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
8. Medical/psychological contraindication to magnetic resonance imaging (MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal toxicity assessed using Common Terminology Criteria for Adverse Events (CTCAE) v5 | 90 days
  Grade 3 or higher gastrointestinal toxicity assessed using Common Terminology Criteria for Adverse Events (CTCAE) v5 within 90 days of completion of radiation therapy

SECONDARY OUTCOMES:
Overall survival | 2 years
  Percentage of patients dying from any cause
Distant progression-free survival | 6 months
  Percentage of patients whose pancreatic cancer does not progress
Patient-reported quality of life (QOL) | 3 and 12 months
  Patient-reported assessments using the National Comprehensive Cancer Network (NCCN) Functional Assessment of Cancer Therapy (FACT) Hepatobiliary Symptom Index, 18-item Hepatobiliary Cancer Subscale (FHSI-18) (NCCN FACT FHSI-18)
  The FACT FHSI-18 is an 18-item scale, each item answered by patients on a scale of 0 ("not at all") to 4 ("very much"). The Total Scale breaks down into 4 subscales as indicated below:
  Total Scale Range: 0-72 (where 72 is good; high scores on each subscale are good)
  Disease-Related Symptoms Subscale-Physical (DRS-P): 12 items, score range 0-48
  Disease-Related Symptoms Subscale - Emotional (DRS-E): 2 items, score range 0-8
  Treatment Side Effects Subscale (TSE): 1 item, score range 0-4
  Function and Well-Being Subscale (FWB): 3 items, score range 0-12
  To view all the FHSI-18 items, see http://www.facit.org/facitorg/questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Parag J Parikh, MD, Principal Investigator — Henry Ford Health System; Percy Lee, MD, Principal Investigator — MD Anderson; Daniel Low, PhD, Principal Investigator — University of California, Los Angeles; Michael Chuong, MD, Principal Investigator — Miami Cancer Institute
Locations (13):
- United States (12):
  - UCLA, Los Angeles, California
  - University of Miami, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health Sciences, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - Cornell University, New York, New York
  - Providence Portland Cancer Center, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Wisconisin, Madison, Wisconsin
- Assuta Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudra S, Jiang N, Rosenberg SA, Olsen JR, Roach MC, Wan L, Portelance L, Mellon EA, Bruynzeel A, Lagerwaard F, Bassetti MF, Parikh PJ, Lee PP. Using adaptive magnetic resonance image-guided radiation therapy for treatment of inoperable pancreatic cancer. Cancer Med. 2019 May;8(5):2123-2132. doi: 10.1002/cam4.2100. Epub 2019 Apr 1. PMID 30932367
- [Derived] Parikh PJ, Lee P, Low DA, Kim J, Mittauer KE, Bassetti MF, Glide-Hurst CK, Raldow AC, Yang Y, Portelance L, Padgett KR, Zaki B, Zhang R, Kim H, Henke LE, Price AT, Mancias JD, Williams CL, Ng J, Pennell R, Pfeffer MR, Levin D, Mueller AC, Mooney KE, Kelly P, Shah AP, Boldrini L, Placidi L, Fuss M, Chuong MD. A Multi-Institutional Phase 2 Trial of Ablative 5-Fraction Stereotactic Magnetic Resonance-Guided On-Table Adaptive Radiation Therapy for Borderline Resectable and Locally Advanced Pancreatic Cancer. Int J Radiat Oncol Biol Phys. 2023 Nov 15;117(4):799-808. doi: 10.1016/j.ijrobp.2023.05.023. Epub 2023 May 19. PMID 37210048
- See also: Parag Parikh, MD: Improving Pancreatic Cancer Survival by using MR Guided Adaptive Radiation — https://vimeo.com/235284105